CLINICAL TRIAL: NCT02474511
Title: the Influence of General Anesthesia on Tumor Metastasis and Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 仁济伦审[2015]058K
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Tumor Recurrence and Metastasis
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Anesthesia, General; Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- general anesthesia: In this group，the patient is received radiofrequency ablation under general anesthesia.
  Interventions: Other: general anesthesia and local anesthesia
- local anesthesia: In this group，the patient is received radiofrequency ablation under local anesthesia.
  Interventions: Other: general anesthesia and local anesthesia

INTERVENTIONS:
Other: general anesthesia and local anesthesia — the patient received generalanesthesia and local anesthesia randomly

SUMMARY:
The purpose of this study was to investigate whether general anesthesia will affect the postoperative recurrence and metastasis of malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III Primary liver cancer tumor is single and diameter is less than 3 centimeter There is no major vascular invasion phenomenon, no lymph nodes or extrahepatic metastases The Child - Pugh belong to type A or type B

Exclusion Criteria:

* Had a history of liver surgery (including radiofrequency ablation) Severe disease of heart, lung, kidney, the immune system INR > 1.5 or platelet count is less than 45000 cells/mm3 History of opioid addiction Metastatic liver tumors Not sure of primary liver cancer Don't agree to participate in this experiment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patient with primary liver cancer.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumor recurrence and metastasis | 3 years
  Follow-up of patients with tumor recurrence and metastasis after Radiofrequency ablation to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China